CLINICAL TRIAL: NCT00211874
Title: Improving Heart Failure Care in Minority Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GCO 99-0347; AHRQ R01 HS10402-01 (Other: AHRQ)
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Congestive Heart Failure (CHF); Systolic Dysfunction
Keywords: Congestive heart failure; nurse management; effectiveness trial; quality improvement; minority communities; disease management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse-management (Experimental): nurse-led intervention focused on specific management problems
  Interventions: Behavioral: Nurse-management
- Usual Care (No Intervention): Usual care as control group

INTERVENTIONS:
Behavioral: Nurse-management — bilingual nurses counseled patients on diet, medication adherence, and self-management of symptoms through an initial visit and regularly scheduled follow-up telephone calls and facilitated evidence-based changes to medications in discussions with patients' clinicians.
  Other Names: Nurse-based disease management
  Arms: Nurse-management

SUMMARY:
For congestive heart failure (CHF) patients with systolic dysfunction, a randomized controlled trial compared nurse-based disease management to address problems in patient and clinician management with usual care for effects on hospitalization and functioning among ethnically-diverse patients in ambulatory practices.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) disproportionately afflicts Black and elderly people, and is a leading cause of hospitalization > 65 years. Although effective therapies can improve functioning and survival in patients with systolic dysfunction, many may not be receiving the full benefit of existing knowledge, including counseling on self-management and appropriate doses of medications. Patients play a critical role in managing a chronic condition such as CHF, but may not have the skills to do so. Clinicians may not provide counseling or medications consistent with evidence-based guidelines.

Systematic reviews of clinical-behavior change have suggested that interventions targeted to specific problems are more likely to be successful. Based on shortfalls identified in patient self-management and clinical care in Harlem, a predominately non-white area in northern Manhattan, we tailored a nurse-management intervention to address the problems documented, and evaluated its effectiveness in a randomized controlled trial. This trial among primarily-minority patients addresses important gaps in this literature: the study targeted problems documented among CHF patients in Harlem, enrolled patients from ambulatory practices, randomly assigned patients between nurse-management and usual care, and evaluated their subsequent health-related outcomes. Hypothesis: the nurse-management program would result in nurse patients' having fewer hospitalizations and reporting better functioning.

ELIGIBILITY:
Inclusion Criteria:

* • adults >18 years,

  * systolic dysfunction documented on a cardiac test (echocardiography, radionuclide ventriculography, myocardial stress sestamibi/thallium testing, or left-heart catheterization),
  * English- or Spanish-speaking,
  * community-dwelling at enrollment, and
  * current patient in a general medicine, geriatrics, or cardiology clinic or office at a participating site.

Exclusion Criteria:

* • medical conditions that prevented a patient's interacting with the nurse, including blindness, deafness, and cognitive impairment;

  * medical conditions that required individualized management that might differ from standard protocol, namely pregnancy, renal dialysis, and terminal illness; and
  * procedures that corrected systolic dysfunction, such as heart transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2000-09; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Short Form 12 questionnaire | 12 months
  self-reported physical functioning as measured by the physical component score on the Short Form 12 questionnaire

SECONDARY OUTCOMES:
Number of hospitalizations | 12 months
  number of hospitalizations in 12 month period
Minnesota Living with Heart Failure Questionnaire | 12 months
  self-reported physical functioning as measured by the physical component score on the Minnesota Living with Heart Failure Questionnaire
Number of deaths | 12 months
  deaths measured by the reporting of death by patient family or recording in the National Death Index

CONTACTS AND LOCATIONS:
Overall Officials: Jane Sisk, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai; Paul Hebert, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - Mount Sinai School of Medicine, New York, New York
  - Metropolitan Hospital, New York, New York
  - North General Hospital, New York, New York
  - Harlem Hospital, New York, New York

REFERENCES:
- [Result] Sisk JE, Hebert PL, Horowitz CR, McLaughlin MA, Wang JJ, Chassin MR. Effects of nurse management on the quality of heart failure care in minority communities: a randomized trial. Ann Intern Med. 2006 Aug 15;145(4):273-83. doi: 10.7326/0003-4819-145-4-200608150-00007. PMID 16908918
- [Result] Horowitz CR, Rein SB, Leventhal H. A story of maladies, misconceptions and mishaps: effective management of heart failure. Soc Sci Med. 2004 Feb;58(3):631-43. doi: 10.1016/s0277-9536(03)00232-6. PMID 14652059
- [Result] Pignone MP, DeWalt DA. Health literacy and heart failure care in minority communities. Ann Intern Med. 2007 Feb 20;146(4):312; author reply 312. doi: 10.7326/0003-4819-146-4-200702200-00014. No abstract available. PMID 17310058